CLINICAL TRIAL: NCT00342108
Title: Cortical Visual Impairment and Visual Attentiveness: The Effect of Visual and Cross-Modal Environments on Children Diagnosed With Cerebral Palsy and Cortical Visual Impairment
Brief Title: Cortical Visual Impairment and Visual Attentiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Amichai Brezner, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4162-AB-CTIL
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Cerebral Palsy; Cortical Visual Impairment
MeSH Terms: conditions — Cerebral Palsy; Blindness, Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Diagnosis: CP, moderate to severe MR and CVI
  Interventions: Behavioral: cross-modal sensory stimulation
- 2 (Experimental): Diagnosis: CP, Moderate to severe MR, no visual impairment
  Interventions: Behavioral: cross-modal sensory stimulation

INTERVENTIONS:
Behavioral: cross-modal sensory stimulation — comparison of participant response to unimodal visual stimulation and to bimodal sensory stimulation

SUMMARY:
This study will investigate the effect of enhanced visual and cross-modal environments upon the visual attentiveness of multiply handicapped children diagnosed with Cerebral Palsy (CP) and Cortical Visual Impairment (CVI).

Research Hypothesis

1. Adapted visual environments which present controlled auditory, tactile, proprioceptive or contrasting visual background stimulation will enhance the visual attentiveness to a given visual stimulus of children diagnosed with CP and CVI.
2. Systematic, repetitive, visual stimulation over time, improves the visual attentiveness and/or visual-motor responses of CP-CVI children.
3. The analysis of additional behavioral responses to visual stimuli is a critical component in evaluating the perceptual development of visual attention in CP-CVI children.

Use of Noldus: The Observer, an advanced objective computerized observation program, will enable precise detection of the neurobehavioral responses of the participants. Both overt and covert responses will be observed, analyzed and correlated to identify the level of attention of each participant.

ELIGIBILITY:
Inclusion Criteria:

* two to twelve years of age
* diagnosis of: CP, mental retardation (MR) and CVI (Control group participants without visual disability)

Exclusion Criteria:

* N/A

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Eye Movements | within the testing session

SECONDARY OUTCOMES:
Other behavioural responses | within the testing session

CONTACTS AND LOCATIONS:
Overall Officials: Amichai Brezner, MD, Principal Investigator — Dept. of Pediatric Rehabilitation Sheba Medical Center Israel
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel